CLINICAL TRIAL: NCT04741204
Title: Metformin Use to Reduce Disparities in Newly Diagnosed Breast Cancer Response to Neoadjuvant Treatment
Brief Title: Metformin Use to Reduce Disparities in Newly Diagnosed Breast Cancer
Acronym: METBC
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Limited staff to carry out study
Sponsor: Woman's (Other)
Collaborators: Our Lady of the Lake Hospital (Other); American Cancer Society, Inc. (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-20-013
Record Dates: First submitted 2021-01-28; First posted 2021-02-05 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer Stage; Insulin Resistance; Racial Bias
Keywords: metformin; breast cancer; racial disparity; tumor regression
MeSH Terms: conditions — Insulin Resistance; Racism; Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Breast cancer tumor response rate to metformin treatment prior to surgery in black vs. white women.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- White women (Experimental): White women on metformin Extended release 750 mg BID
  Interventions: Drug: Metformin Extended Release Oral Tablet
- Black women (Experimental): Black women on metformin Extended release 750 mg BID
  Interventions: Drug: Metformin Extended Release Oral Tablet

INTERVENTIONS:
Drug: Metformin Extended Release Oral Tablet — initial dose of metformin of 750 mg Q.D. (with dinner) for 3-4 weeks. They then will be increased to the final dose of 750 mg BID (breakfast and dinner) until the end of the study.
  Other Names: metformin XR; metformin ER

SUMMARY:
Breast cancer is one of the most common malignancies in women globally, with ~1.4 million new cases diagnosed annually Breast cancer is one of the leading causes of cancer-related morbidity and mortality among women worldwide. While diabetes/insulin-resistance and breast cancer are distinct diseases, insulin-signaling plays a central role in both illnesses. Insulin activates key cancer processes including epithelial-mesenchymal transition (EMT), tissue inﬂammation, motility, and angiogenesis. There are key opportunities to impact and prevent hyperinsulinemia during breast cancer prevention, surgical assessment, and chemotherapy. Given the high prevalence of undiagnosed pre-diabetes and diabetes in the United States and worldwide, preoperative screening to identify such patients prior to surgical intervention is warranted. While it is not standard of care to test for insulin-resistance during the course of breast cancer screening and treatment, it is standard of care to screen and test high risk women for insulin-resistance as part of whole woman care. Given the important role insulin signaling plays in driving signaling pathways that promote aggressive cancer biology, more attention should be paid by cancer physicians to screening and treating insulin resistance. Several studies have reinforced a link between breast cancer risk and diabetes. Moreover, metformin significantly reduces breast cancer risk, compared to patients who are not using metformin and is independent of diabetes status. As metformin has an association with decreased breast cancer recurrence, as well as potentially improved survival, disparities in insulin resistance between black and white women with breast cancer is important to investigate. It is hypothesized that metformin decreases the development of resistance in breast cancer cells, thereby allowing current chemotherapy agents to work synergistically with metformin. Our objective is to elucidate whether or not metformin is efficacious in improving insulin resistance in black and white women with breast cancer and if racial disparities in breast cancer prognosis can be partially explained by differences in pre-diagnosis insulin resistance which are improved with metformin therapy.

DETAILED DESCRIPTION:
Even as cancer research has led to more advanced, targeted cancer treatments than ever before, not all patients are able to reap the benefits of these efforts, as demonstrated by their persistently worse survival outcomes, lack of accrual onto clinical trials, and lower rates of genetic testing. According to the American Cancer Society, black patients have the highest death rates and shortest duration of survival of any racial or ethnic group in the U.S. for most cancers. Black individuals with cancer are 25% more likely to die of their disease than white patients. Although persisting across tumor types, this disparity is particularly evident among black women, whose population-based breast cancer mortality rate is higher than white women. Compared with white women, black women have a 42% higher breast cancer mortality rate and twofold higher incidence of biologically aggressive triple-negative disease. Additionally, the American Cancer Society reported that black women are significantly more likely to die of breast cancer than white women, a disparity that has increased over time.

For decades, researchers attributed higher mortality rates to socioeconomic factors such as inadequate health insurance, fewer years of education and lower income. However, research now supports the hypothesis that tumor biologic differences among black women could have a greater impact on response to treatment and outcomes. Some disparities are a function of environmental stressors influenced by race that affect biology. Body mass index (BMI), obesity, and rates of diabetes are higher for African Americans. Obesity is associated with a 35% to 40% increased risk of breast cancer recurrence and death and therefore poorer survival outcomes. This association is most clearly established for estrogen receptor-positive breast cancer, with the relationship in triple-negative and human epidermal growth factor receptor 2-overexpressing subtypes less well established. A range of biologic mechanisms that may underlie this association has been identified. In an early meta-analysis evaluating BMI and breast cancer risk, the authors found that every 5 kg/m2 increase of BMI was associated with 12% increased risk of breast cancer in postmenopausal women. The inflammatory and endocrine effects of obesity, a major risk factor for type 2 diabetes (T2DM), have been proposed as central mechanisms explaining associations between diabetes and cancer.

Approximately ~ 10% of all cancers in women are attributable at least in part to obesity, with certain tumor types exhibiting an even stronger relationship between excess weight and cancer risk. Among these are breast and colon cancer, in which obesity promotes tumor appearance, progression, and metastasis in rodent models and in human patients. Obesity is associated with elevated insulin levels and increased insulin resistance. Insulin, a member of a family of growth factors that includes insulin-like growth factor (IGF)-I and IGF-II, exerts mitogenic effects on normal and malignant breast epithelial cells, acting via insulin and IGF-I receptors. Insulin resistance could lead to compensatory hyperinsulinemia, which enhances the cross-binding of insulin to the insulin-like growth factor-1 (IGF-1) receptors expressed on breast epithelial cells. Moreover, hyperinsulinemia may also accelerate the pathogenesis of breast cancer by stimulation of hepatic IGF-1 synthesis and inhibition the hepatic expression of IGF-1 receptors, leading to an increased circulating IGF-1 level. Interfering with insulin signaling may slow tumor growth while activation of the insulin receptor may promote tumor progression.

Hyperinsulinemia, which occurs as a consequence of lipid-induced insulin resistance and may also hasten its progression, is one of many putative links that may explain the association between obesity and cancer. Insulin promotes tumor cell division in vitro and plasma insulin concentrations are independently correlated with an increased risk and accelerated progression of both breast and colon cancer. High levels of fasting insulin identify women with poor outcomes in whom more effective treatment strategies should be explored. Black women are twice as likely to have prediabetes and type 2 diabetes as white women; improved monitoring of blood sugar and insulin levels to identify women with prediabetes could provide opportunities for reduction of the incidence of ER-negative breast cancer. A 12-week to 18-week course of chemotherapy appears to statistically significantly increase metabolic syndrome (MetS) and related anthropometrics, biomarkers of glucose metabolism, and inflammation in patients with early-stage breast cancer with no preexisting MetS. Lifestyle interventions such as diet and exercise may be preventive approaches for use during chemotherapy to reduce the onset of MetS in patients with breast cancer.

Breast cancer (BC) is one of the most common malignancies occurring in females. Weight loss and lifestyle interventions, as well as metformin and other obesity-targeted therapies, are promising avenues that require further study in women with breast cancer. The oral insulin-sensitizing drug metformin is a first line therapeutic in the management of T2DM. Metformin is a biguanide agent that reduces hepatic glucose production, increases hepatic fatty acid oxidation, reduces inflammation, and improves peripheral insulin sensitivity These activities reduce circulating glucose and insulin levels, although the exact mechanisms by which metformin achieves these effects are not well understood. In prior clinical studies elevated insulin levels were associated with poorer outcomes in patients with breast cancer; the use of metformin in women with early-stage breast cancer has been shown to reduce insulin levels. Metformin may affect breast cancer proliferation depending on a woman's insulin resistance, with decreased proliferation occurring in women with an increased homeostasis model assessment index (more insulin resistant). The rate of pathologic complete response was three time higher in women receiving neoadjuvant treatment for early-stage breast cancer plus metformin than in those women receiving neoadjuvant therapy without metformin.. Metformin has also been shown to have antiproliferative activity in vitro against multiple cancer cells lines. An early meta-analysis performed on T2DM patients taking metformin with cancer reported a 31% reduction in the incidence of new cancers including pancreas, colorectal, breast, and lung. Recent meta-analyses confirm that individuals with T2DM who also have lung, colorectal, and liver cancer derive significant survival benefits regarding clinical outcomes if also on metformin. Patients with breast cancer benefited from metformin treatment in terms of all cause survival (overall survival or chance of remaining alive after diagnosis). Data from previously conducted studies has shown metformin decreased the incidence of cancer and cancer-related deaths in patients with diabetes. Cellular glucose metabolism is linked tightly with the proliferation and development of breast cancer. Several studies suggested that metformin reduces the incidence of breast cancer in T2DM patients. Cancer cells show enhanced glucose uptake and metabolism and prefer glycolysis over OXPHOS, which is called the "Warburg effect." The noted specialty of metformin is to decrease glucose levels, thereby limiting the availability of energy for cancer cells. Metformin was also shown to decrease FAS expression, an essential component of the fatty acid synthesis pathway, thus affecting the survival of cancer cells. Metformin affects AMP-activated protein kinase, which effects mitochondrial energy generation and may deprive malignant, inefficient cells of energy and therefore reduce their potential growth rate. Although some of the observations [with metformin] imply not just [preventing] a progression of cancer but an incidence of cancer, which might suggest broader effects than merely energy deprivation. In parallel with that data, there are experimental findings that support a direct effect of metformin on specific pathways that mediate or promote cancer. It's been shown in both animal models and cell lines that metformin can inhibit some of the key steps that are important for tumors to grow, such as promotion of cell growth, motility, invasion, and migration. These findings provide us with new insight in the use of metformin combined with other drugs to treat tumors.

Epidemiologic studies suggest that metformin use may be associated with both reduced cancer incidence and mortality. In a study, Tesneg and colleagues analyzed data from 493,704 men and 502,139 women without colon cancer covered by national health insurance from 2003 to 2005, assessing whether metformin use had a protective effect. Although patients with diabetes had a higher risk for developing colon cancer, patients assigned metformin had a 27% reduced risk, according to researchers. Comparing patients with diabetes for less than 1 year, between 1 and 2 years, and at least 3 years with patients without diabetes, adjusted RRs were 1.308 (95% CI, 1.02-1.679), 1.087 (95% CI, 0.9-1.313) and 1.185 (95% CI, 1.055-1.33), respectively. The duration of metformin use showed an inverse trend, according to researchers, with an RR of 0.643 (95% CI, 0.49-0.845) in users for at least 3 years vs. nonusers. A few mechanisms have been hypothesized to explain what may be happening. The most prominent theory is the idea that metformin activates a specific protein kinase, which down regulates the mTOR signaling pathway, which is important for tumor cell metabolism. More broadly, there is some evidence that insulin itself - and insulin-related pathways - may promote cancers. There is the thought that metformin does modulate insulin and sensitizes cells to insulin, and that may also have something to do with its effects. Our objective is to elucidate whether or not metformin is efficacious in improving insulin resistance in black and white women with breast cancer and if racial disparities in breast cancer prognosis can be partially explained by differences in pre-diagnosis insulin resistance which are improved with metformin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic white or black females
* Age > = 18 years
* English speaking
* Newly diagnosed breast cancer
* BMI > = 25 (must be overweight)
* Insulin-resistant (as determined by 2 hour 75 gm oral glucose tolerance test (OGTT)). Concentrations and trajectories of insulin and glucose at 0, 30, 60, and 120 min during an oral glucose tolerance test will undergo mathematical modeling. The numbers for defining insulin resistance have been established in the Woman's Laboratory and are interpreted by the pathologists.

Exclusion Criteria:

* Metastatic Disease
* Current diagnosis of Diabetes or diagnosed with diabetes (as determined by HbA1C> 6.5)
* Having surgery prior to chemotherapy
* Medical conditions for which metformin is contraindicated (gastrointestinal and renal failure),
* Abnormal CBC (defined by a baseline platelet count of less than 130 and a baseline absolute neutrophil count of less than 1000). In addition, baseline hemoglobin of less than 10, if there is no evidence of a concurrent nutritional deficiency (like iron). [Patients simply needing something like iron to correct the anemia will not be excluded].

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — genetic XX
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Tumor progression | 6 to 12 months
  breast cancer response rate to metformin treatment prior to surgery pathologic response to treatment at surgery will be defined by the following categories: 0-no response; 1-partial response; and 2-complete response with metformin therapy

SECONDARY OUTCOMES:
Fasting glucose levels | 6 to 12 months
  Fasting glucose at start of OGTT
Mean glucose stimulated levels after an OGTT | 6 to 12 months
  Mean blood glucose (MBG) concentrations will be calculated by summing glucose values obtained at 0, 30, 60, and 120 minutes during the OGTT and dividing by 4.
Homeostatic Model Assessment of Insulin Resistance Index (HOMA-IR) | 6 to 12 months
  HOMA will be calculated using the equation: fasting insulin concentration (μIU/mL) × fasting glucose concentration (mmol/L) 22.5
Matsuda's insulin sensitivity index (SIOGTT) | 6 to 12 months
  SIOGTT will be calculated according to the formula:
  10,000/√ [fasting glucose (mg/dL) ×fasting insulin (μU/L) × [MPG × MSI during OGTT], where MPG (mg/dL) is mean plasma glucose OGTT, and MSI (μIU/mL) is mean serum insulin during OGTT
Early pancreatic β-cell response | 6 to 12 months
  IGI/HOMA-IR estimated as the insulinogenic index (IGI) derived from the ratio of the increment of insulin to that of glucose 30 minutes after a glucose load (insulin 30 min - insulin 0 min/glucose 30 min - glucose 0 min) corrected for by the relative level of insulin resistance
Insulin secretion-sensitivity index (ISSI) | 6 to 12 months
  IS-SI derived by applying the concept of the disposition index to measurements obtained during the 2-h OGTT and calculated as the index of insulin secretion factored by insulin resistance (ΔINS/ΔPG 30 x Matsuda SIOGTT) during the OGTT

OTHER OUTCOMES:
Recurrence rate of breast cancer | 3 years
  follow-up for recurrence of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ericka Seidemann, MA, Study Chair — Woman's Hospital, Louisiana; Cynthia Harper-Weinstein, Study Chair — Mary Bird Perkins Cancer center
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No